CLINICAL TRIAL: NCT05778266
Title: Effect of L-citrulline and HIIT on Arterial Stiffness, Body Composition, and Lipid Profile in Adolescents with Steatosis Associated with Metabolic Dysfunction (MASLD)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad de Guanajuato (Other)
Responsible Party: Principal Investigator, Ma Eugenia Garay Sevilla, Titular Research Professor, Universidad de Guanajuato
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PWV-MAFLD-HIIT-CITRULLINE
Record Dates: First submitted 2023-02-19; First posted 2023-03-21 (Actual); Last update posted 2024-12-20 (Actual); Status verified 2023-03

CONDITIONS: Metabolic Dysfunction-Associated Fatty Liver Disease; Obesity, Adolescent; Arterial Stiffness
Keywords: MAFLD; Obesity; Adolescents; PWV; AIx75; HIIT; L-citrulline supplementation
MeSH Terms: conditions — Pediatric Obesity; Obesity | interventions — Citrulline; Carboxymethylcellulose Sodium

STUDY DESIGN:
Intervention Model Description: An intervention with exercise in modality of High-Intensity Interval Training (HIIT) and Oral administration of L-citrulline (L-cit) or placebo (Pl) as follows:
  Group L-cit + HIIT: capsules of 6 g of citrulline will be supplemented per day, distributed as 3 g (4 capsules) in the morning before the first meal and 3 g in the evening before sleep for a period of 12 weeks. The sessions of HIIT will be made 3 days per week in a stationary bicycle Group Pl + HIIT: Carboxymethyl cellulose will be used as placebo. 4 capsules will be taken in the morning before the first meal and 4 capsules at night before going to sleep for a period of 12 weeks. The sessions of HIIT will be made 3 days per week in a stationary bicycle.
  Group L-cit without HIIT: capsules of citrulline will be supplemented per day, distributed as 3 g (4 capsules) in the morning before the first meal and 3 g (4 capsules) in the evening before sleep for a period of 12 weeks. This group will not made exercise.
Who Masked: Participant, Investigator
Masking Description: The selection of which group each adolescent will belong to, will be made by randomization by computer numbers by a researcher from the department of medical sciences of the University of Guanajuato, who is not involved in treatment and follow-up. The researcher will designated into a placebo or L-cit group. The investigator and the participants will not know the group which they belong.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- L-Cit + HIIT (Active Comparator): adolescents will be supplemented with 6 g/day of L-citrulline and 3 sessions per week of HIIT for 12 weeks
  Interventions: Dietary Supplement: L-citrulline; Other: High Intensity Intervals Training
- L-Cit (Active Comparator): adolescents will be supplemented with 6 g/day of L-citrulline but without do exercise for 12 weeks
  Interventions: Dietary Supplement: L-citrulline
- Placebo + HIIT (Placebo Comparator): adolescents will be supplemented with 6 g/day of Carboxymethyl cellulose and 3 sessions per week of HIIT for 12 weeks
  Interventions: Dietary Supplement: Carboxymethyl cellulose; Other: High Intensity Intervals Training

INTERVENTIONS:
Dietary Supplement: L-citrulline — oral supplementation of pure L-citrulline (6 g) for twelve weeks
  Arms: L-Cit; L-Cit + HIIT
Dietary Supplement: Carboxymethyl cellulose — oral supplementation of Carboxymethyl cellulose (6 g) as a placebo, for twelve weeks
  Other Names: Placebo
  Arms: Placebo + HIIT
Other: High Intensity Intervals Training — participants will have sessions 3 days a week for twelve weeks
  Other Names: HIIT
  Arms: L-Cit + HIIT; Placebo + HIIT

SUMMARY:
Obesity and metabolic dysfunction-associated steatotic liver disease (MASLD) accelerate the appearance of arterial stiffness due to inflammatory and oxidative stress mechanisms producing increased vascular tone and increasing the risk of cardiovascular disease. This arterial stiffness can be measured through pulse wave velocity (PWV). Obesity and MAFLD have multifactorial components, high fructose diet and sedentary lifestyle are causing the onset of these diseases earlier in life such as in adolescence. L-citrulline, a non-protein amino acid, has shown positive effects on improving nitric oxide synthesis which improves endothelial function, as well as results on the metabolic profile in MASLD. High intensity interval training (HIIT) has also shown benefits on endothelial function improving the metabolic profile of people with obesity and MASLD with the advantage of decreasing the time required to perform the physical activity. A clinical study will be conducted with 45 adolescents (15-19 years old) with MASLD and the participants will be divided into 3 groups to perform HIIT and supplement with citrulline or placebo for 12 weeks.

DETAILED DESCRIPTION:
The investigators hypothesize that citrulline and HIIT have additive effects on endothelial function in people with obesity and MASLD, in addition to improving metabolic, lipid and hepatic steatosis profile. the researcher´s aim is to evaluate the effect of citrulline and HIIT on arterial stiffness assessed by PWV in adolescents with MASLD. For this the investigators will perform a randomized, double-blind clinical study in 45 adolescents with MASLD and obesity, who will be supplemented with 6 g per day with L-citrulline or placebo (Carboxymethylcellulose) and will perform HIIT sessions for 12 weeks. At the beginning and at the end of the intervention, the level of arterial stiffness by means of PWV, body composition, biochemical and metabolic data, as well as the degree of hepatic steatosis will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of obesity and metabolic associated-dysfunction steatotic liver disease associated with (MASLD) and with moderate or severe steatosis
* History of physical inactivity
* They should not be under treatment with any dietary supplement or polyvitamins for weight loss at least 6 months before the study.
* They should not be smokers.
* Not have a diagnosis of any chronic degenerative disease
* Adolescents without fracture or musculoskeletal injury
* Patients without surgical procedures at least 1 month prior to the protocol.
* Women who are not pregnant or use oral contraceptives

Exclusion Criteria:

* Participants who do not complete at least 80% of the training sessions.
* Participants who miss 2 consecutive weeks of training.
* Who do not ingest the L-citrulline supplement or placebo.
* Participants who present allergy or intolerance to L-citrulline.
* Participants who present any injury during the intervention period that prevents them from performing the training.

Ages: 15 Years to 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 43 (Actual)
Dates: Start 2023-03-14 (Actual); Primary Completion 2024-01-15 (Actual); Study Completion 2024-04-30 (Actual)

PRIMARY OUTCOMES:
Arterial Stiffness | 12 weeks
  The degree of arterial stiffness will be evaluated by oscillometric device (Mobil-O Graph). This device assesses Pulse Wave Velocity
Reflected Wave | 12 weeks
  The Augmentation Index (AIx) measures the percentage of the pressure increase that is caused by the premature arrival of the reflected wave and is expressed as the ratio of PAo and PP multiplied by 100. AIx@75 is AIx corrected to a heart rate of 75 beats per minute. The Mobil-O Graph device also evaluates AIx@75
Degree of hepatic steatosis | 12 weeks
  The degree of hepatic steatosis will be evaluated by abdominal ultrasound. It will be diagnosed as:
  1. Moderate, when sound attenuation is added.
  2. Severe, when the wall of the portal vessels and the diaphragm are not visible.

SECONDARY OUTCOMES:
Glucose metabolism: glucose | 12 weeks
  Glucose will be evaluated by the Lakeside glucose oxidase method (GOD-PAPTM).
Glycated hemoglobin (HbA1c) | 12 weeks
  Glycated hemoglobin (HbA1c) will be measured by reflectance spectrophotometry, by boronic acid affinity.
Insuline Resistance | 12 weeks
  Insulin level will be measured by ELISA (ALPCO) method. The Homeostatic Model Assessment Index (HOMA-IR) will be calculated to determine insulin resistance.
Lipid profile | 12 weeks
  The lipid profile will be measured by the modified Huang method.
VO2max | 12 weeks
  VO2max is a measure of aerobic exercise capacity. It will be performed on a cycloergometer. Every 2 minutes 0.5 kp will be increased and HR will be measured minute by minute with a portable monitor (Polar HO1). When the participant no longer maintains the 60 rpm cadence or reaches the maximum perceived exertion on the modified Borg scale (9 or 10), the test is terminated.
Arterial Pressure | 12 weeks
  Is pressure exerted by the blood on the artery wall. The mobil-O Graph also evaluates arterial pressure and reports it as Dyastolic Pressure (DAP), Systolic Pressure (SAP) and Mean Arterial Pressure (MAP)
Body composition | 12 weeks
  Bioelectrical impedance will be used to assess total body composition as fat free mass (FFM), fat mass (FM) and total body water, using the standard configuration.
  The portable, multi-frequency In body S10 device will be used and it reports body composition in percentage (%)

CONTACTS AND LOCATIONS:
Overall Officials: Ma. Eugenia Garay-Sevilla, PhD, Principal Investigator — Universidad de Guanajuato; Alan Arturo Rodriguez-Carrillo, Bachelor, Study Chair — Universidad de Guanajuato
Locations (1):
- Universidad de Guanajuato, León, Guanajuato, Mexico

IPD SHARING:
Plan to Share IPD: No
At the request of the researcher

REFERENCES:
- [Derived] Rodriguez-Carrillo AA, Espinoza-Vargas MR, Vargas-Ortiz K, Ibarra-Reynoso LDR, Olvera-Juarez M, Gomez-Ojeda A, Garay-Sevilla ME, Figueroa A. Impact of L-Citrulline Supplementation and HIIT on Lipid Profile, Arterial Stiffness, and Fat Mass in Obese Adolescents with Metabolic-Dysfunction-Associated Fatty Liver Disease: A Randomized Clinical Trial. Nutrients. 2025 Jan 23;17(3):402. doi: 10.3390/nu17030402. PMID 39940261